CLINICAL TRIAL: NCT03809806
Title: Four-arm Mesh for Vaginal Stump Prolapse: Surgical Technique and Outcomes
Brief Title: Four-arm Mesh for Vaginal Stump Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Paweł Miotła, Clinical Professor, Medical University of Lublin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02/2019
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Pelvic Organ Prolapse; Sexual Function Abnormal
Keywords: vaginal stump prolapse; sexual function; quality of life
MeSH Terms: conditions — Pelvic Organ Prolapse; Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: Patients with vaginal stump prolapse who had undergone hysterectomy in the past
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients after hysterectomy (Other): modified anterior transvaginal mesh surgery
  Interventions: Procedure: 4-arm polypropylene mesh surgery; Diagnostic Test: The Female Sexual Function Index (FSFI) questionnaire; Diagnostic Test: King Health Questionnaire (KHQ); Diagnostic Test: Pelvic Organ Prolapse Quantification (POPQ) staging; Diagnostic Test: Postoperative questionnaire; Diagnostic Test: The Short Form Health Survey (SF 36) questionnaire

INTERVENTIONS:
Procedure: 4-arm polypropylene mesh surgery — Pelvic reconstructive procedures were performed with the use of 4-arm mesh:upper arms through- anterior part of obturator foramens, lower arms-ischiorectal fossas and sacrospinal ligaments.
Diagnostic Test: The Female Sexual Function Index (FSFI) questionnaire — patients fulfilled questionnaire before and 1 year after procedure
Diagnostic Test: King Health Questionnaire (KHQ) — patients fulfilled questionnaire before and 1 year after procedure
Diagnostic Test: Pelvic Organ Prolapse Quantification (POPQ) staging — Pelvic Organ Prolapse staging before and 1 year after the procedure
Diagnostic Test: Postoperative questionnaire — Postoperative questionnaire assessing quality of life fulfilled by patients 1 year after procedure
Diagnostic Test: The Short Form Health Survey (SF 36) questionnaire — patients fulfilled questionnaire before and 1 year after procedure

SUMMARY:
To estimate the safety and efficacy of performing modified anterior transvaginal mesh surgery using polypropylene mesh for treatment of advanced urogenital prolapse after hysterectomy (stage III and IV vc Pelvic Organ Prolapse Quantification [POP-Q] system staging).

DETAILED DESCRIPTION:
Pelvic reconstructive procedures were primarily performed using the transvaginal four arm polypropylene mesh, which was inserted through: upper arms- anterior part of obturator foramens, lower arms-ischiorectal fossas and sacrospinal ligaments. All patients underwent hysterectomy in the past apart from one which underwent vaginal hysterectomy during the procedure. Perineoplasty was performed additionally, if indicated. Subjective and objective evaluations included Pelvic Organ Prolapse Quantification [POP-Q] staging, preoperative and 1-year postoperative questionnaires were performed.

ELIGIBILITY:
Inclusion Criteria:

* Pelvic Organ Prolapse Quantification (POPQ) III and IV vc after hysterectomy

Exclusion Criteria:

* malignant diseases
* unability to understand informed consent

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Pelvic Organ Prolapse Quantification (POPQ) 1 year after procedure | 1 year
  assessment of POPQ 1 year after mesh operation, Pelvic Organ Prolapse Quantification system (POP-Q) refers to an objective, site-specific system for describing, quantifying, and staging pelvic support in women. It provides a standardized tool for documenting, comparing, and communicating clinical findings with proven interobserver and intraobserver reliability

SECONDARY OUTCOMES:
Sexual function 1 year after procedure | 1 year
  assessment of sexual function before and 1 year after the procedure with the use of The Female Sexual Function Index questionnaire
Urinary incontinence 1 year after procedure | 1 year
  assessment of urinary incontinence before and 1 year after the procedure with the use of the Urogenital Distress Inventory (UDI 6) and the Incontinence Impact Questionnaire (IIQ 7) questionnaire
quality of life 1 year after procedure | 1 year
  assessment of quality of life before and 1 year after the procedure with the use of The Short Form Health Survey (SF 36)

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Rechberger, Professor, Principal Investigator — 2nd Gynecology Department Medical University in Lublin
Locations (1):
- 2nd Gynecology Department, Lublin, Poland

IPD SHARING:
Plan to Share IPD: No